CLINICAL TRIAL: NCT04669106
Title: Mineral and Enzyme Deficiency Diseases Associated With Nutritional Diseases in Society
Status: Completed | Type: Observational
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, DINA KEUMALA SARI, Principal Investigator, Universitas Sumatera Utara
Other Study IDs: USumateraUtara 3
Record Dates: First submitted 2020-11-26; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Nutrient Deficiency
Keywords: nutritional deficiency; macronutrient; mineral; enzyme; stunting
MeSH Terms: conditions — Malnutrition; Calcinosis; Growth Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy group: 90 research subjects coming from mothers who had healthy children
  Interventions: Other: laboratory clinical trial study
- Stunting group: 90 research subjects came from mothers who had stunted children or other nutritional disorders
  Interventions: Other: laboratory clinical trial study

INTERVENTIONS:
Other: laboratory clinical trial study — The research stage consisted of two stages, the first stage was the initial screening of the primary data of the research subjects, namely by analyzing food intake including mineral intake data, the diet of the research subjects, mineral and enzyme levels, and data on soil conditions in the area. The second stage was to analyze the relationship between the existing variables so that the most significant relationship was seen between the differences in diet, mineral content, enzyme levels, and soil content between the two groups.

SUMMARY:
Nutritional deficiency disease is a disease caused by nutritional deficiencies, including macronutrients and micronutrients. Macronutrient diseases are diseases caused by deficiency of protein, fat and carbohydrates. This deficiency will usually show clinical symptoms that directly affect nutritional status. This study aims to study and examine mineral intake, dietary patterns of research subjects, mineral and enzyme levels, and soil condition data. The number of research subjects to be taken was 180 subjects with 90 research subjects coming from mothers who had healthy children and 90 research subjects came from mothers who had stunted children or other nutritional disorders. The research stage will run after going through the inclusion of research subjects, namely mothers who have healthy children and mothers who have nutritionally deficient children, aged 20-40 years. The research stage consisted of two stages. The statistical analysis used is to use the ANOVA test, which will then compile a manuscript.

DETAILED DESCRIPTION:
This study aims to study and examine mineral intake, dietary patterns of research subjects, mineral and enzyme levels, and soil condition data. The number of research subjects to be taken was 180 subjects with 90 research subjects coming from mothers who had healthy children and 90 research subjects came from mothers who had stunted children or other nutritional disorders. The research stage will run after going through the inclusion of research subjects, namely mothers who have healthy children and mothers who have nutritionally deficient children, aged 20-40 years. The research stage consisted of two stages. The statistical analysis used is to use the ANOVA test, which will then compile a manuscript.

This research is a case control study, with primary data collection, is a laboratory clinical trial study on the subject of mothers who have children aged 2-3 years, aged 20-40 years. The number of research subjects to be taken was 180 subjects with 90 research subjects coming from mothers who had healthy children and 90 research subjects came from mothers who had stunted children or other nutritional disorders.

The research stage consisted of two stages, the first stage was the initial screening of the primary data of the research subjects, namely by analyzing food intake including mineral intake data, the diet of the research subjects, mineral and enzyme levels, and data on soil conditions in the area. The second stage was to analyze the relationship between the existing variables so that the most significant relationship was seen between the differences in diet, mineral content, enzyme levels, and soil content between the two groups. The statistical analysis used was to use the ANOVA test.

ELIGIBILITY:
Inclusion Criteria:

* mothers who had healthy children

Exclusion Criteria:

* mothers who have healthy children and mothers who have nutritionally deficient children

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: The number of research subjects to be taken was 180 subjects with 90 research subjects coming from mothers who had healthy children and 90 research subjects came from mothers who had stunted children or other nutritional disorders. The research stage will run after going through the inclusion of research subjects, namely mothers who have healthy children and mothers who have nutritionally deficient children, aged 20-40 years.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
calsium, vitamin D, zinc and ferrum serum level | up to 1 day
  calsium, vitamin D, zinc and ferrum serum level in the mother's blood
lipase and amylase enzime pacreatic serum level | up to 1 day
  lipase and amylase enzime pacreatic serum level in the mother's blood
dietary intake per day | up to 2 day
  dietary intake per day of mother and child

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Universitas Sumatera Utara, Medan, North Sumatra, Indonesia

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT04669106/Prot_ICF_000.pdf